CLINICAL TRIAL: NCT05199636
Title: Effect of Dragon Fruit Consumption on Glycaemic Response and Blood Pressure in Individuals at Risk of Type 2 Diabetes
Brief Title: Effect of Dragon Fruit Consumption in Individuals at Risk of Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford Brookes University (Other)
Responsible Party: Principal Investigator, Dr. Sangeetha Thondre, Senior Lecturer, Oxford Brookes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UREC 211527
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Blood Pressure; Glucose Intolerance
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dragon fruit product (Experimental): A dragon fruit beverage
  Interventions: Other: Dragon fruit product
- General health advice (No Intervention): Based on Eatwell guide and guidelines for type 2 diabetes prevention from the National Institute for Health and Care Excellence (NICE)

INTERVENTIONS:
Other: Dragon fruit product — Frozen dragon fruit based beverage
  Arms: Dragon fruit product

SUMMARY:
In this project, an edible product based on dragon fruit will be tested to determine its effect on blood glucose levels and blood pressure in individuals at risk of type 2 diabetes. The effect of a product from dragon fruit on fasting plasma glucose and blood pressure will be assessed by a parallel study design with two groups and 16 participants in each one. Secondary outcomes such as inflammation biomarkers, lipid profile and oxidative stress markers also will be determined in blood samples.

DETAILED DESCRIPTION:
This will be a parallel study in which two different treatments will be evaluated to determine their effect on glucose, blood pressure, and other outcomes including dietary assessment in individuals at risk of diabetes. The study will last 4 weeks and will involve 3 testing sessions. The participants (N=32) will be randomly divided into two groups and asked either to consume daily a dragon fruit based beverage or to follow a general health guidelines for 4 weeks. The treatment will be taken once a day and a 24 hours dietary recall will be recorded three times during the intervention; the results provided will contribute to understanding the role of polyphenols from the edible products based on dragon fruit on glucose metabolism, blood pressure and linked biomarkers.

Treatment for testing group 1, will include an advice that involve following general health guidelines based on Eatwell Guide and guidelines for type 2 diabetes prevention from the National Institute for Health and Care Excellence (NICE) for 4 weeks. Treatment for testing group 2, will involve drinking a dragon fruit based beverage daily for 4 weeks.

The first visit will start by asking participants to take part in a 24 hours dietary recall and by recording anthropometric measurements. Blood pressure will be taken after 10 minutes of rest (three measurements at five minutes intervals). Venous blood sample will be taken by venepunture to determine fasting blood glucose and biomarkers. Then a standard glucose drink (75g of glucose in 250 ml of water) will be given to determine glucose tolerance, a further venous sample will be taken after 2 hours. Between the 2 hours, finger-prick blood samples will be taken at 0, 15, 30, 45, 60, 90 and 120 minutes intervals, to evaluate the glycaemic and insulin response profile. The treatment will be given to the participant to start the intervention.

The second session will be held 2 weeks after the treatment begins and the protocol established above for the first session will be followed.

After 4 weeks of treatment the third session will be conducted, as mentioned in first and second sessions. Anthropometric measurements will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-50 years who fulfil at least two of the following inclusion criteria:

  * Have a first grade relative with diabetes (parent, brother, or sister)
  * Have a BMI ≥ 25.0.
  * Have a sedentary lifestyle.

Exclusion Criteria:

* • Covid-19 related symptoms, during the last 7 days.

  * Allergies to dragon fruit.
  * Diabetes, hypertension, or renal disease.
  * Medication that requires prescription.
  * Pregnant or breastfeeding.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Blood glucose response | 2 hours
  Blood glucose in venous blood sample
Blood pressure | 15 minutes
  Systolic and diastolic blood pressure

SECONDARY OUTCOMES:
Plasma insulin response | 2 hours
  Insulin response in fingerprick blood sample
C-reactive protein | 5 minutes
  C-reactive protein
HbA1C | 5 minutes
  Glycated hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Sangeetha Thondre, PhD, Principal Investigator — Oxford Brookes University
Locations (1):
- Oxford Brookes Centre for Nutrition and Health, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flores-Verastegui MIM, Coe S, Tammam J, Almahjoubi H, Bridle R, Bi S, Thondre PS. Effects of Frozen Red Dragon Fruit Consumption on Metabolic Markers in Healthy Subjects and Individuals at Risk of Type 2 Diabetes. Nutrients. 2025 Jan 25;17(3):441. doi: 10.3390/nu17030441. PMID 39940297